CLINICAL TRIAL: NCT00577863
Title: B3D-MC-GHDF: Community Experience of Subjects With Osteoporosis Using the Forteo B Pen to Self Administer Once Daily Teriparatide Therapy
Brief Title: Study of the Experience of Patients With Osteoporosis Using the Forteo B Pen to Self Administer Once Daily Teriparatide Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10586; B3D-MC-GHDF
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2009-06-24 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: teriparatide — Subcutaneous injection of teriparatide 20 micrograms once daily using the Forteo B Pen. The primary phase of the study is 8 weeks after which time patients may participate in a study extension until the patient completes their maximum duration of teriparatide therapy or the Forteo B Pen becomes commercially available.
  Other Names: LY333334

SUMMARY:
This study is being conducted to collect information from subjects with osteoporosis regarding their experience using the Forteo B Pen to self-administer teriparatide in the community setting. Information collected during this study will be used to assess the need for changes to the Forteo B-Pen User Manual and patient educational tools. Additionally, the information generated from patients during this trial will be reviewed to assess the acceptability of the Forteo B Pen for commercial launch.

ELIGIBILITY:
Inclusion Criteria:

1. Men with primary or hypogonadal osteoporosis or postmenopausal women with osteoporosis in the opinion of the investigator. Subjects must be at high risk for fracture in the opinion of the investigator.
2. Willing to be trained and use the pen-injector daily to the satisfaction of study site personnel.
3. Able to read, understand, and respond to self-administered questionnaires.
4. Without language barrier, cooperative, and expected to return for all follow-up procedures.
5. Have provided written informed consent to participate in this study, according to local regulations after being informed of the risks, medications, and procedures to be used in the study.

   Exclusion Criteria:
6. Any disease of sufficient severity to preclude treatment with teriparatide or participation in and completion of the study as defined by the investigator.
7. Having laboratory values, such as elevated serum calcium, precluding teriparatide treatment as defined by the investigator.
8. Subjects who have an increased baseline risk of osteosarcoma, including those with: Paget's disease of the bone or unexplained elevations of alkaline phosphatase, children and young adults with open epiphyses, and subjects who have received external beam or implant radiation therapy involving the skeleton.
9. History of malignant neoplasms in the 5 years prior to study entry, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated, or history of carcinoma in situ of the cervix or uterus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montgomery, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beckley, West Virginia

REFERENCES:
- [Derived] Dore RK, Feldman RG, Taylor KA, See K, Dalsky GP, Warner MR. Patient experience with a new teriparatide delivery device. Curr Med Res Opin. 2009 Oct;25(10):2413-22. doi: 10.1185/03007990903173074. PMID 19656016
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are reported for participants who received at least one injection of study drug.
Groups:
- Current Users: A Current User was defined as a patient with ≥8 weeks experience with the original delivery device (Forteo 1.1 Pen), including uninterrupted use during the 4 weeks prior to enrollment. Patients received teriparatide 20 mcg/day during the study using the Forteo B Pen.
- Not Current Users: A Not Current User could be either treatment naïve or have experience with the original device (Forteo 1.1 Pen) that did not meet the criteria outlined for a Current User. Thus, a Not Current User could have used the original delivery device for up to 22 months, as long as they had not used the original device within 4 weeks of enrollment. Patients received teriparatide 20 mcg/day during the study using the Forteo B Pen.
Period: Overall Study
Arm/Group | Current Users | Not Current Users
Started | 92 | 108
Received at Least One Injection | 92 | 107
Completed | 82 | 94
Not Completed | 10 | 14
Not completed — Adverse Event | 4 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Entry Criteria Exclusion | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Sponsor Decision | 2 | 7
Not completed — Did Not Receive at Least One Injection | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Current Users | Not Current Users | Total
Number analyzed (Participants) | 92 | 107 | 199
Age Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.01) | 68.5 (11.54) | 67.9 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 96 | 178
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 92 | 107 | 199
Previous Teriparatide Use [Number; unit: participants]
  Yes | 92 | 27 | 119
  No | 0 | 80 | 80
Race/Ethnicity [Number; unit: participants]
  Caucasian | 87 | 104 | 191
  African | 0 | 1 | 1
  Hispanic | 2 | 1 | 3
  East Asian | 3 | 1 | 4
Duration of Prior Forteo 1.1 Pen Experience [Mean (Standard Deviation); unit: weeks] | 36.5 (23.01) | 12.9 (16.33) | 31.2 (23.78)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Forteo B Pen Complaints at 8 Weeks
Description: Summary of number of complaints, and common complaints (at least 3% complaint rate), from subjects using Forteo B Pen. Functional Complaints were related to device malfunction; Nonfunctional were related to either cosmetic or perception concerns.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug.
Measure: Number; unit: number of complaints
Groups:
- Forteo B Pen Users: All subjects using the Forteo B Pen to self-administer teriparatide in the community setting for 8 weeks.
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 199
number of complaints
  All Complaints | 47
  Complaint Category: Functional | 4
  Complaint Category: Nonfunctional | 27
  Nonfunctional (4%): Pen too large, awkward, bulky | 8
  Complaint Category: User Manual Related | 16
  User Manual (3.5%): No information on alcohol swab | 7

2. Secondary Outcome: Summary of Subject Preference Assessments - Overall Preference
Description: To assess overall subject preferences for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: All participants who received at least one injection of study drug and are currently using the Forteo 1.1 Pen who answered the question.
Measure: Number; unit: participants
Groups:
- Forteo 1.1 Pen Users: Current users of the Forteo 1.1 Pen.
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 2
  2 | 1
  3 = No Preference | 4
  4 | 6
  5 = Strong Preference for Forteo B Pen | 79

3. Secondary Outcome: Summary of Subject Preference Assessments - Learning to Use the Pen
Description: To assess subject preferences for learning to use the pen for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 2
  2 | 0
  3 = No Preference | 8
  4 | 7
  5 = Strong Preference for Forteo B Pen | 75

4. Primary Outcome: Number of Subjects With Forteo B Pen Complaints at 8 Weeks
Description: Number of subjects with complaints after 8 weeks, and common complaints (at least 3% complaint rate), using Forteo B Pen. Functional Complaints were related to device malfunction; Nonfunctional were related to either cosmetic or perception concerns.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug.
Measure: Number; unit: number of participants with complaints
Groups:
- Forteo B Pen Users: All subjects using the Forteo B Pen to self-administer teriparatide in the community setting for 46 weeks.
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 199
number of participants with complaints
  All Complaints | 31
  Complaint Category: Functional | 4
  Complaint Category: Nonfunctional | 19
  Nonfunctional (4%): Pen too large, awkward, bulky | 8
  Complaint Category: User Manual Related | 14
  User Manual (3.5%): No information on alcohol swab | 7

5. Secondary Outcome: Summary of Subject Preference Assessments - Attaching a New Needle
Description: To assess subject preferences for attaching a new needle for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 2
  2 | 0
  3 = No Preference | 36
  4 | 8
  5 = Strong Preference for Forteo B Pen | 46

6. Secondary Outcome: Summary of Subject Preference Assessments - Setting the Dose
Description: To assess subject preferences for setting the dose for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 2
  2 | 0
  3 = No Preference | 3
  4 | 8
  5 = Strong Preference for Forteo B Pen | 79

7. Secondary Outcome: Summary of Subject Preference Assessments - Injecting a Dose
Description: To assess subject preferences for injecting a dose for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 2
  2 | 1
  3 = No Preference | 16
  4 | 6
  5 = Strong Preference for Forteo B Pen | 67

8. Secondary Outcome: Summary of Subject Preference Assessments - Force on the Plunger Needed to Inject a Dose
Description: To assess subject preferences for force on the plunger needed to inject a dose for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 2
  2 | 3
  3 = No Preference | 14
  4 | 11
  5 = Strong Preference for Forteo B Pen | 62

9. Secondary Outcome: Summary of Subject Preference Assessments - Assurance That Drug is Delivered
Description: To assess subject preferences for assurance that drug is delivered for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 4
  2 | 3
  3 = No Preference | 23
  4 | 16
  5 = Strong Preference for Forteo B Pen | 46

10. Secondary Outcome: Summary of Subject Preference Assessments - Removing a Used Needle
Description: To assess subject preferences for removing a used needle for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 3
  2 | 1
  3 = No Preference | 36
  4 | 7
  5 = Strong Preference for Forteo B Pen | 45

11. Secondary Outcome: Summary of Subject Preference Assessments - Overall Ease of Use
Description: To assess subject preferences for overall ease of use for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 1
  2 | 3
  3 = No Preference | 4
  4 | 3
  5 = Strong Preference for Forteo B Pen | 81

12. Secondary Outcome: Summary of Subject Preference Assessments - Use of the User Manual/Instructions for Use That Came With the Pen
Description: To assess subject preferences for use of the User Manual/Instructions for Use that came with the pen for the Forteo 1.1 Pen or the Forteo B Pen through a questionnaire at Visit 2 completed by subjects who switch from the Forteo 1.1 Pen prior to the study entry to the Forteo B Pen during study participation.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Forteo 1.1 Pen Users
Number analyzed (Participants) | 92
participants
  1 = Strong Preference for Forteo 1.1 Pen | 3
  2 | 2
  3 = No Preference | 15
  4 | 9
  5 = Strong Preference for Forteo B Pen | 63

13. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Remove Pen From Package
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to remove the pen from the package.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 0
  3 | 5
  4 | 19
  5 = Strongly Agree | 174

14. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Read Label
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to read the label.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 2
  3 | 6
  4 | 25
  5 = Strongly Agree | 165

15. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Learn to Use the Pen
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to learn to use the pen.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 1
  2 | 1
  3 | 0
  4 | 16
  5 = Strongly Agree | 180

16. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Remove The Pen Cap
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to remove the pen cap.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 0
  3 | 1
  4 | 15
  5 = Strongly Agree | 182

17. Secondary Outcome: Summary of Subject Perception (Attibutes) Assessments - Easy to Replace The Pen Cap
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to replace the pen cap.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 0
  3 | 0
  4 | 14
  5 = Strongly Agree | 184

18. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Attach a New Needle
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to attach a new needle.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 1
  2 | 0
  3 | 5
  4 | 17
  5 = Strongly Agree | 175

19. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Remove a Used Needle
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to remove a used needle.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 197
participants
  1 = Strongly Disagree | 0
  2 | 2
  3 | 9
  4 | 18
  5 = Strongly Agree | 168

20. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Set the Dose
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to set the dose.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 197
participants
  1 = Strongly Disagree | 1
  2 | 1
  3 | 3
  4 | 9
  5 = Strongly Agree | 183

21. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Push the Black Injections Button to Administer the Dose
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to push the black injections button to administer the dose.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 0
  3 | 4
  4 | 19
  5 = Strongly Agree | 175

22. Secondary Outcome: Summary of Subject Perceptions (Attributes) Assessments - Easy to Hold the Pen While Injecting
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to hold the pen while injecting.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 2
  3 | 8
  4 | 29
  5 = Strongly Agree | 159

23. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Easy to Use the Forteo B Pen Instructions For Use
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how easy it was to use the Forteo B Pen Instructions for Use.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 0
  3 | 8
  4 | 16
  5 = Strongly Agree | 174

24. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Overall Ease of Use
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of the overall ease of use.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 0
  3 | 1
  4 | 18
  5 = Strongly Agree | 179

25. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - To What Extent Are You Satisfied With the Forteo B Pen
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how satisfied they were with the Forteo B Pen.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Very Dissatisfied | 0
  2 | 0
  3 | 4
  4 | 18
  5 = Very Satisfied | 176

26. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - How Confident Are You That You Receive the Medication With Your Forteo B Pen
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how confident they were that they received the medication with the Forteo B Pen.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 197
participants
  1 = Not At All Confident | 2
  2 | 4
  3 | 10
  4 | 32
  5 = Very Confident | 149

27. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Convenient for Me to Use
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of how convenient Forteo B Pen was to use.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 1
  3 | 1
  4 | 19
  5 = Strongly Agree | 177

28. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Reduces My Reluctance to Take Injections
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of whether the Forteo B Pen reduces their reluctance to take injections.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 197
participants
  1 = Strongly Disagree | 3
  2 | 2
  3 | 14
  4 | 27
  5 = Strongly Agree | 151

29. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Helps Me Manage My Osteoporosis At Home
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of whether the Forteo B Pen helps them manage their osteoporosis when they are at home.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  1 = Strongly Disagree | 0
  2 | 1
  3 | 3
  4 | 15
  5 = Strongly Agree | 179

30. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Helps Me Manage My Osteoporosis Away From Home
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of whether the Forteo B Pen helps them manage their osteoporosis when they are away from home.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 194
participants
  1 = Strongly Disagree | 2
  2 | 5
  3 | 19
  4 | 26
  5 = Strongly Agree | 142

31. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - Reusing Needles
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject response on whether or not they sometimes reuse needles.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  No | 197
  Yes - Occasionally | 0
  Yes - Often | 0
  Yes - Rarely | 1

32. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - When Do You Attach a Needle
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject response on when they attach a needle to their Forteo B Pen.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 199
participants
  Immediately Before Each Injection | 197
  Several Hours Before Each Use | 2
  At Home If Injection Is Completed Away From Home | 5
  Other | 0

33. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - When Do You Remove the Needle
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject response on when they remove the needle from their Forteo B Pen.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 198
participants
  Immediately | 197
  When I Get Home If Injection Completed Away | 0
  Other | 1

34. Secondary Outcome: Summary of Subject Perception (Attributes) Assessments - What Could Be Done to Improve the Forteo B Pen Instructions For Use
Description: To assess overall subject perception of the device performance and acceptability through a questionnaire completed by all subjects at Visit 3. Subject perception of what could be done to improve the Forteo B Pen Instructions for Use.
Time Frame: 8 weeks
Population: All participants who received at least one injection of study drug and who answered the question.
Measure: Number; unit: participants
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 199
participants
  Larger Print | 22
  More Color | 5
  Less Color | 1
  More Pictures | 7
  Less Pictures | 3
  More Detail in the Description | 10
  Less Detail in the Description | 1
  More Questions and Answers | 11
  No Improvements Needed | 156

35. Primary Outcome: Summary of Forteo B Pen Complaints at 46 Weeks
Description: as for outcome 1
Time Frame: 46 weeks
Population: All participants who received at least one injection of study drug.
Measure: Number; unit: number of complaints
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 199
number of complaints
  All Complaints | 58
  Complaint Category: Functional | 9
  Functional (3%): Stopped working, wouldn't inject | 6
  Complaint Category: Nonfunctional | 32
  Nonfunctional (4%): Pen too large, awkward, bulky | 8
  Complaint Category: User Manual Related | 17
  User Manual (3.5%): No information on alcohol swab | 7

36. Primary Outcome: Number of Subjects With Forteo B Pen Complaints at 46 Weeks
Description: Number of subjects with complaints after 46 weeks, and common complaints (at least 3% complaint rate), using Forteo B Pen. Functional Complaints were related to device malfunction; Nonfunctional were related to either cosmetic or perception concerns.
Time Frame: 46 weeks
Population: All participants who received at least one injection of study drug.
Measure: Number; unit: number of participants with complaints
Arm/Group | Forteo B Pen Users
Number analyzed (Participants) | 199
number of participants with complaints
  All Complaints | 37
  Complaint Category: Functional | 9
  Functional (3%): Stopped working, wouldn't inject | 6
  Complaint Category: Nonfunctional | 21
  Nonfunctional (4%): Pen too large, awkward, bulky | 8
  Complaint Category: User Manual Related | 14
  User Manual (3.5%): No information on alcohol swab | 7

ADVERSE EVENTS:
Groups:
- Teriparatide: Teriparatide 20 micrograms per day
Arm/Group | Teriparatide
Serious Adverse Events (participants affected / at risk) | 14
Other Adverse Events (participants affected / at risk) | 134
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Teriparatide
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1/199 (1)
Arrhythmia (Cardiac disorders) | 1/199 (1)
Atrial fibrillation (Cardiac disorders) | 1/199 (1)
Bradycardia (Cardiac disorders) | 1/199 (1)
Cardiac failure congestive (Cardiac disorders) | 1/199 (1)
Cardiogenic shock/Death (Cardiac disorders) | 1/199 (1)
Diarrhoea (Gastrointestinal disorders) | 1/199 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1/199 (1)
Pneumonia (Infections and infestations) | 1/199 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1/199 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1/199 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1/199 (1)
Dehydration (Metabolism and nutrition disorders) | 1/199 (1)
Fluid overload (Metabolism and nutrition disorders) | 1/199 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/199 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/199 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/199 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/199 (1)
Syncope (Nervous system disorders) | 1/199 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/199 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Teriparatide
Anaemia (Blood and lymphatic system disorders) | 4/199 (4)
Ear pain (Ear and labyrinth disorders) | 2/199 (2)
Vertigo (Ear and labyrinth disorders) | 2/199 (2)
Abdominal pain (Gastrointestinal disorders) | 2/199 (2)
Gastritis (Gastrointestinal disorders) | 2/199 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4/199 (4)
Nausea (Gastrointestinal disorders) | 8/199 (8)
Vomiting (Gastrointestinal disorders) | 3/199 (3)
Fatigue (General disorders) | 9/199 (9)
Injection site bruising (General disorders) | 2/199 (2)
Injection site haemorrhage (General disorders) | 2/199 (2)
Non-cardiac chest pain (General disorders) | 2/199 (2)
Oedema peripheral (General disorders) | 4/199 (4)
Drug hypersensitivity (Immune system disorders) | 2/199 (2)
Bronchitis (Infections and infestations) | 5/199 (5)
Gastroenteritis viral (Infections and infestations) | 3/199 (3)
Helicobacter infection (Infections and infestations) | 2/199 (2)
Influenza (Infections and infestations) | 4/199 (4)
Nasopharyngitis (Infections and infestations) | 4/199 (4)
Pneumonia (Infections and infestations) | 2/199 (2)
Sinusitis (Infections and infestations) | 7/199 (7)
Upper respiratory tract infection (Infections and infestations) | 12/199 (13)
Urinary tract infection (Infections and infestations) | 8/199 (10)
Back injury (Injury, poisoning and procedural complications) | 2/199 (2)
Contusion (Injury, poisoning and procedural complications) | 8/199 (9)
Excoriation (Injury, poisoning and procedural complications) | 2/199 (3)
Fall (Injury, poisoning and procedural complications) | 2/199 (2)
Joint sprain (Injury, poisoning and procedural complications) | 2/199 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2/199 (2)
Colonoscopy (Investigations) | 2/199 (2)
Heart rate irregular (Investigations) | 2/199 (2)
Vitamin D decreased (Investigations) | 2/199 (2)
Weight decreased (Investigations) | 3/199 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 2/199 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2/199 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2/199 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9/199 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8/199 (8)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2/199 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3/199 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7/199 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 3/199 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5/199 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/199 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2/199 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2/199 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3/199 (3)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 2/199 (2)
Dizziness (Nervous system disorders) | 8/199 (8)
Headache (Nervous system disorders) | 6/199 (6)
Tremor (Nervous system disorders) | 2/199 (2)
Depression (Psychiatric disorders) | 4/199 (4)
Insomnia (Psychiatric disorders) | 2/199 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3/199 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/199 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2/199 (2)
Rash (Skin and subcutaneous tissue disorders) | 4/199 (6)
Dental prosthesis placement (Surgical and medical procedures) | 2/199 (2)
Joint arthroplasty (Surgical and medical procedures) | 2/199 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days